CLINICAL TRIAL: NCT06362941
Title: A Single-Center Prospective Evaluation of an Oral Hair Supplement to Improve Hair Strength and Support Growth in Women and Men with Self-Perceived Hair Thinning
Brief Title: Evaluation of an Oral Hair Supplement to Improve Hair Strength and Support Growth in Women and Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nutraceutical Wellness Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NW-HGN-01
Record Dates: First submitted 2024-04-08; First posted 2024-04-12 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2024-09

CONDITIONS: Hair Thinning
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Intervention Model Description: Single Group Assignment 6-month, single-center, prospective interventional study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Nutrafol Hair Growth Supplement (Experimental): 5 commercially available hair growth nutraceuticals will be evaluated. Treatment groups will be assigned according to the investigator's discretion. Efficacy comparisons will not be made across treatment groups.
  Interventions: Dietary Supplement: Nutrafol Women's Hair Growth Supplemnt; Dietary Supplement: Nutrafol Women's Balance Hair Growth Supplement; Dietary Supplement: Nutrafol Women's Vegan Hair Growth Supplement; Dietary Supplement: Nutrafol Women's Postpartum Hair Growth Supplement; Dietary Supplement: Nutrafol Men's Hair Growth Supplement

INTERVENTIONS:
Dietary Supplement: Nutrafol Women's Hair Growth Supplemnt — Hair growth supplement for women ages 18 - 44.
Dietary Supplement: Nutrafol Women's Balance Hair Growth Supplement — Hair growth supplement for women ages 45 - 70.
Dietary Supplement: Nutrafol Women's Vegan Hair Growth Supplement — Hair growth supplement for women ages 18 - 44. This treatment group may also include subjects who do not follow a plant-based diet for purposes of extending the product claims beyond the initially studied demographic of women primarily adhering to a plant-based diet.
Dietary Supplement: Nutrafol Women's Postpartum Hair Growth Supplement — Hair growth supplement for women ages 18 - 44. This product will be studied in the general women population and not postpartum women.
Dietary Supplement: Nutrafol Men's Hair Growth Supplement — Hair growth supplement for men ages 25 - 50.

SUMMARY:
A single-center, open-label, prospective study to demonstrate the efficacy of an oral supplement to improve the strength and support the growth of thinning hair in men and women with self-perceived hair thinning.

DETAILED DESCRIPTION:
Female and male subjects will be enrolled in this single-site, open-label, prospective, interventional study evaluating 5 treatment regimens to improve the appearance of thinning hair. All treatment regimens are commercially available nutraceutical hair growth supplements. 50 subjects will be enrolled into each of the 5 supplement groups. Subjects will undergo a baseline, 90 day, and 180 day visit and will have compliance phone calls at Days 45 and 135. Study assessments will include a dermatologist investigator hair assessment, a hair pull test, light microscope hair shaft diameter assessment, and a subject questionnaire.

ELIGIBILITY:
Inclusion Criteria:

1. Female or male subjects with concerns and/or signs of hair thinning.
2. The subjects must meet the age characteristics based on their supplement group assignment.
3. Subjects are Fitzpatrick Skin Types I to VI.
4. Subjects must be in good general health.
5. Subjects must be classified with thinning hair by the study dermatologist.
6. Willing to maintain the same hair length, hairstyle, and coloring practices for the duration of the study. Subjects who have color-treated hair must have the color treatment performed at the same time interval prior to each visit.
7. Willing to use a mild non-medicated shampoo and conditioner for the duration of the study (medicated shampoo and conditioner refer to any prescription shampoo or conditioner as well as any over-the counter medicated shampoo or conditioner, such as those for treatment of dandruff or promoting hair growth).
8. Willing and able to adhere to the same dietary lifestyles for the duration of the study
9. Subjects must express willingness to cooperate with the investigator and comply to study requirements.
10. Subjects must demonstrate the ability to read and understand all the items in the informed consent document.
11. Subjects must agree not to use any other hair supplements or start a new vitamin supplement during the study.
12. Subject has signed an Informed Consent Form in compliance with 21CFR Part 50: "Protection of Human Subjects."
13. Subject is dependable and able to follow directions and is willing to comply with the schedule of visits.

Exclusion Criteria:

1. Any previous or current acute or chronic medical or hair condition, which in the investigator's opinion, may interfere with the study results or increase the study participation risks to the subject.
2. Subjects possessing signs of severe female or male pattern hair loss or alopecia (including androgenetic and traction alopecia) as determined by the study dermatologist.
3. Scalp hair loss on the treatment area, due to disease, injury, or medical therapy
4. Subjects who are not willing to use only the assigned oral study supplement and no new oral supplements during the study.
5. Subjects who have demonstrated a previous hypersensitivity reaction to any of the ingredients of the study product.
6. Subjects, who are pregnant, breast feeding, or planning a pregnancy.
7. Subjects with clinically significant unstable medical disorders.
8. Subjects who are unwilling or unable to comply with the requirements of the protocol.
9. Subjects who have history of a psychological illness or condition that would interfere with their ability to understand and/or follow the requirements of the study.
10. Subjects with any planned surgeries and/or invasive medical procedures during the course of the study.
11. History of surgical correction of hair loss on the scalp (i.e., hair transplant).
12. Use of any products or devices purported to promote scalp hair growth (e.g., finasteride or minoxidil) within the 6 months prior to the Baseline Visit.
13. Females who have recently (within the last 6 months) started the use of hormones for birth control or hormone replacement therapy (HRT). Women currently using Scalp hair loss on the treatment area, due to disease, injury, or medical therapy
14. hormones for birth control or HRT must have been on a stable dose (6 months or longer) in order to be eligible for the study (the initiation of HRT or birth control should not have been associated with the initiation of hair loss/thinning).
15. History of burning, flaking, itching, and stinging of the scalp.
16. Utilization of low-level lasers for hair growth in the last three months.
17. Known history or recent blood work indicating iron deficiency, bleeding disorders or platelet dysfunction syndrome as well as subjects receiving anticoagulant therapy or smokers with usage >20 cigarettes/day.
18. Use of any medications or medicated shampoos that are known to potentially cause hair loss or affect hair growth, as determined by the Investigator or qualified sub-investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2024-05-20 (Actual); Primary Completion 2025-02-18 (Actual); Study Completion 2025-02-18 (Actual)

PRIMARY OUTCOMES:
Change in hair shaft diameter compared to baseline at Day 180. | 180 days
  The ability of an oral supplement to improve hair shaft strength as evidenced by change in hair shaft diameter from baseline at Day 180 in new scalp hair growth as viewed by the study dermatologist under a light microscope in men and women with self-perceived thinning hair.
Change in hair shaft diameter compared to baseline at Day 90. | 90 days
  The ability of an oral supplement to improve hair shaft strength as evidenced by change in hair shaft diameter from baseline at Day 90 in new scalp hair growth as viewed by the study dermatologist under a light microscope in men and women with self-perceived thinning hair.

SECONDARY OUTCOMES:
Change in broken hairs recovered from the hair pull test compared to baseline at Day 180 | 180 days
  The ability of an oral supplement to improve hair strength as evidenced by a change in the number of broken hairs recovered from the hair pull test at Day 180 compared to baseline in men and women with self-perceived thinning hair.
Change in broken hairs recovered from the hair pull test compared to baseline at Day 90 | 90 days
  The ability of an oral supplement to improve hair strength as evidenced by a change in the number of broken hairs recovered from the hair pull test at Day 90 compared to baseline in men and women with self-perceived thinning hair.
Change in hair breakage during the hair pull test compared to baseline at Day 180 | 180 Days
  The ability of an oral supplement to promote longer hair as evidenced by change in hair breakage observed in the hair pull test compared to baseline at Day 180.
Change in hair breakage during the hair pull test compared to baseline at Day 90 | 90 Days
  The ability of an oral supplement to promote longer hair as evidenced by change in hair breakage observed in the hair pull test compared to baseline at Day 90.
Change in the number of hairs recovered from the hair pull test compared to baseline at Day 180 | 180 Days
  The ability of an oral supplement to improve hair shedding as evidenced by a change in the number of hairs recovered from the hair pull test compared to baseline at Day 180 in men and women with self-perceived thinning hair.
Change in the number of hairs recovered from the hair pull test compared to baseline at Day 90 | 90 Days
  The ability of an oral supplement to improve hair shedding as evidenced by a change in the number of hairs recovered from the hair pull test compared to baseline at Day 90 in men and women with self-perceived thinning hair.
Subject Self-Perceived Improvement in Hair Quality at Day 180 | 180 Days
  The ability of an oral supplement to improve hair growth and quality in men and women with self-perceived thinning hair as measured by self-assessment questionnaires using a 5-point ordinal scale (0=excellent, 1=good, 2=average, 3=poor, 4=very poor) at Day 180.
Subject Self-Perceived Improvement in Hair Quality at Day 90 | 90 Days
  The ability of an oral supplement to improve hair growth and quality in men and women with self-perceived thinning hair as measured by self-assessment questionnaires using a 5-point ordinal scale (0=excellent, 1=good, 2=average, 3=poor, 4=very poor) at Day 90.

CONTACTS AND LOCATIONS:
Locations (1):
- Dermatology Consulting Services, High Point, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Draelos Z, Farris PK, Hazan A, Raymond I. A 6-Month, Prospective, Multi-arm Study for the Efficacy of Standardized Nutraceuticals to Improve Hair Fiber Thickness and Strength. Dermatol Ther (Heidelb). 2025 Oct 31. doi: 10.1007/s13555-025-01582-0. Online ahead of print. PMID 41171588